CLINICAL TRIAL: NCT02209480
Title: Randomized Controlled Trial on the Efficacy of F.M. Alexander Technique in Chronic Neck Pain Patients
Brief Title: Alexander Technique Neck Pain
Acronym: ATNeck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principle Investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-3497
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Chronic Non-specific Neck Pain
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alexander Technique (Experimental): 5 lessons of AT, each lasting up to 45 minutes, weekly intervals The lessons aimed at sensory awareness of everyday movements and movement sequences, such as sitting, walking, lying, or lifting in order to replace habitual patterns using conscious control; and different techniques were applied, such as demonstration, verbal instructions, hands on techniques and others
  Interventions: Behavioral: Alexander Technique
- Heat pad application (Active Comparator): 5 treatments by means of a heat pad, 15-0 minutes, sitting or lying position, quiet room Heat pad: Zapp-Sack® contained certain grains and a ginger extract, and could be heated up in the microwave.
  Interventions: Device: Heat pad application
- guided imagery (Active Comparator): guided imagery relaxation technique , 45 minutes, 5 sessions in weekly rhythm including body scan, breathing relaxation, visualization
  Interventions: Behavioral: guided imagery

INTERVENTIONS:
Behavioral: Alexander Technique
  Arms: Alexander Technique
Device: Heat pad application
  Arms: Heat pad application
Behavioral: guided imagery
  Arms: guided imagery

SUMMARY:
This study aimed to test the efficacy of five Alexander Technique lessons compared to the same period of heat pad application and guided imagery in patients with chronic non-specific neck pain.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* chronic non-specific neck pain
* at least 3 months
* 40mm pain intensity on visual analog scale

Exclusion Criteria:

* neck pain as consequence of disc protrusion or prolapse, whiplash, congenital deformity of the spine, spinal stenosis, neoplasm, inflammatory rheumatic disease, neurological disorder,
* active oncologic disease
* affective disorder
* addiction
* psychosis.
* pregnancy
* invasive treatment of the spine within the previous three weeks
* spinal surgery
* previous experiences in Alexander Technique
* ongoing application for disability pension
* simultaneous participation in other clinical trials on neck pain

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
neck pain intensity | 5 weeks
  neck pain intensity measured on a 100mm visual analog scales
  1. comparison Alexander technique vs. heat pad
  2. comparison Alexander technique vs. guided imagery

SECONDARY OUTCOMES:
quality of life | 5 weeks
  quality of life measured by the SF-36 questionnaire
Pain on motion | 5 weeks
  pain on motion (movement of head in different directions) measured by the POM (Lauche, 2014, pain medicine)
Medication | 5 weeks
  weekly dose of medication calculated as the defined daily dose according to WHO
functional disability | 5 weeks
  measured by the neck disability index (NDI)
satisfaction | 5 weeks
  satisfaction measured on a visual analog scale and via questions like "would you consider using it again" or "would you recommend it"
safety | 5 weeks
  any adverse event during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany

REFERENCES:
- [Result] Lauche R, Schuth M, Schwickert M, Ludtke R, Musial F, Michalsen A, Dobos G, Choi KE. Efficacy of the Alexander Technique in treating chronic non-specific neck pain: a randomized controlled trial. Clin Rehabil. 2016 Mar;30(3):247-58. doi: 10.1177/0269215515578699. Epub 2015 Mar 31. PMID 25834276